CLINICAL TRIAL: NCT01237613
Title: Prospective Study on Artelon® Tissue Reinforcement in Repair of Chronic Ruptures and Re-ruptures of the Achilles Tendon
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsoring company declared bankrupty
Sponsor: Orthopedic Foot and Ankle Center, Ohio (Other)
Collaborators: Artimplant AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KP027ext
Record Dates: First submitted 2010-09-16; First posted 2010-11-09 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-06

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles; Rupture; Tendon; Artelon
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Artelon (Experimental): This is an open, prospective study with an anticipated enrollment of 10 patients with chronic or repeat Achilles tendon rupture undergoing surgical repair augmented with Artelon® Tissue Reinforcement.
  Interventions: Device: Artelon

INTERVENTIONS:
Device: Artelon — Artelon Tissue Reinforcement

SUMMARY:
The aim of this study is to evaluate the surgical and clinical outcome of Artelon® Tissue Reinforcement in repair of chronic ruptures or re-ruptures of the Achilles tendon, with regard to lower leg and foot function, pain and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a clinically confirmed isolated chronic rupture or rerupture of the Achilles tendon.
2. The patient has been informed about the study and signed the patient consent form.
3. The patient reads, understands and is able to complete the study questionnaires in English.

Exclusion Criteria:

1. The patient has an ongoing infection of the soft tissues of the ankle.
2. The patient has evidence of severe ankle arthritis.
3. The patient has a multi-system or multi-limb trauma.
4. The patient has a major medical condition that would affect quality of life and influence the results of the study.
5. The patient is pregnant
6. The patient is not expected to complete the study according to the investigation plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terrence M Philbin, DO, Principal Investigator — Orthopedic Foot and Ankle Center
Locations (1):
- Orthopedic Foot and Ankle Center, Westerville, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Artelon: This was an open, prospective study with an anticipated enrollment of 10 patients with chronic or repeat Achilles tendon rupture undergoing surgical repair augmented with Artelon® Tissue Reinforcement.
  Artelon: Artelon Tissue Reinforcement
Period: Overall Study
Arm/Group | Artelon
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Artelon
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 54 [38 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: The Foot Function Index (FFI) for Evaluation of Foot Pain and Disability
Time Frame: 3 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Groups:
- Open: This was an open, prospective study with an anticipated enrollment of 10 patients with chronic or repeat Achilles tendon rupture undergoing surgical repair augmented with Artelon® Tissue Reinforcement.
  Artelon: Artelon Tissue Reinforcement
Arm/Group | Open
Number analyzed (Participants) | 0

2. Primary Outcome: The Foot Function Index (FFI) for Evaluation of Foot Pain and Disability
Time Frame: 6 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

3. Primary Outcome: The Foot Function Index (FFI) for Evaluation of Foot Pain and Disability
Time Frame: 12 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

4. Secondary Outcome: The American Orthopaedic Foot and Ankle Society (AOFAS) Clinical Rating System for Ankle-hindfoot
Time Frame: 3 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

5. Secondary Outcome: General Measure of Health-related Quality of Life Using the EuroQoL (EQ-5D) Questionnaire
Time Frame: 3 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

6. Secondary Outcome: Range of Motion, Strength and Calf Circumference
Time Frame: 3 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

7. Secondary Outcome: Subjective Evaluation of Treatment
Time Frame: 3 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

8. Secondary Outcome: Return to Work and Previous Physical Activities
Time Frame: 3 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

9. Secondary Outcome: Clinical Evaluation Including Adverse Events
Time Frame: 3 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

10. Secondary Outcome: The American Orthopaedic Foot and Ankle Society (AOFAS) Clinical Rating System for Ankle-hindfoot
Time Frame: 6 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

11. Secondary Outcome: General Measure of Health-related Quality of Life Using the EuroQoL (EQ-5D) Questionnaire
Time Frame: 6 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

12. Secondary Outcome: Range of Motion, Strength and Calf Circumference
Time Frame: 6 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

13. Secondary Outcome: Subjective Evaluation of Treatment
Time Frame: 6 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

14. Secondary Outcome: Return to Work and Previous Physical Activities
Time Frame: 6 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

15. Secondary Outcome: Clinical Evaluation Including Adverse Events
Time Frame: 6 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

16. Secondary Outcome: The American Orthopaedic Foot and Ankle Society (AOFAS) Clinical Rating System for Ankle-hindfoot
Time Frame: 12 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

17. Secondary Outcome: General Measure of Health-related Quality of Life Using the EuroQoL (EQ-5D) Questionnaire
Time Frame: 12 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Groups:
- Open: This was an open, prospective study with an anticipated enrollment of 10 patientschronic or repeat Achilles tendon rupture undergoing surgical repair augmented with Artelon® Tissue Reinforcement.
  Artelon: Artelon Tissue Reinforcement
Arm/Group | Open
Number analyzed (Participants) | 0

18. Secondary Outcome: Range of Motion, Strength and Calf Circumference
Time Frame: 12 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

19. Secondary Outcome: Subjective Evaluation of Treatment
Time Frame: 12 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

20. Secondary Outcome: Return to Work and Previous Physical Activities
Time Frame: 12 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

21. Secondary Outcome: Clinical Evaluation Including Adverse Events
Time Frame: 12 months
Population: Data not analyzed as study was terminated due to sponsor bankruptcy.
Arm/Group | Open
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Artelon
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artelon (N=4)
Sinusitis (Immune system disorders) | 1 (1)
C-difficile (Gastrointestinal disorders) | 1 (1)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased tenderness over left peroneal and posterior tibial tendons (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The sample size is small due to the study being terminated early because of sponsor bankrupty,

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less